CLINICAL TRIAL: NCT00001469
Title: Genetic Analysis of Hereditary Prostate Cancer
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950158; 95-HG-0158
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Genotyping; Linkage Analysis; Adenocarcinoma; Micro Satellite; Hereditary; Prostate Cancer (hereditary)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Prostate cancer, familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Specimens: Specimens

SUMMARY:
Molecular approaches to the understanding of human neoplastic disease have revealed that multiple genetic alterations are an essential component of tumorigenesis. Both germline and somatic genetic alterations can be involved in the malignant transformation of normal cells. Identification of the genes involved in neoplastic transformation has been approached through the molecular analysis of sporadic cancers and the genetic study of families with an inherited predisposition for cancer. The interplay of these two approaches has led to the characterization of genes such as the retinoblastoma (Rb) gene, the p53 gene and the adenomatous polyposis coli (APC) gene that are all involved in the development of both hereditary and non-hereditary forms of cancer. Inherited mutations in such genes predispose affected families to hereditary cancer syndromes, affording an opportunity to identify genetic lesions that also cause the more common sporadic cancers.

Prostate cancer (PRCA) is the most common cancer diagnosed (1999 estimate 179,300 cases) and the second leading cause of cancer mortality (1999 estimate 37,000 deaths) in men in the United States. Family history is the single strongest risk factor currently known for prostate cancer. This raises the possibility that heritable genetic factors may be involved in the development of this disease in a subset of men. The genetic contribution to diseases of complex origin such as cancer is often most salient in families of early onset cases. Therefore, prostate cancer inheritance following a simple Mendelian pattern may be identified in the families of probands with early-onset cases. Common susceptibility alleles of small effect may be detectable in families with later-onsent and/or less strong family history of PRCA or in case-control data.

DETAILED DESCRIPTION:
Molecular approaches to the understanding of human neoplastic disease have revealed that multiple genetic alterations are an essential component of tumorigenesis. Both germline and somatic genetic alterations can be involved in the malignant transformation of normal cells. Identification of the genes involved in neoplastic transformation has been approached through the molecular analysis of sporadic cancers and the genetic study of families with an inherited predisposition for cancer. The interplay of these two approaches has led to the characterization of genes such as the retinoblastoma (Rb) gene, the p53 gene and the adenomatous polyposis coli (APC) gene that are all involved in the development of both hereditary and non-hereditary forms of cancer. Inherited mutations in such genes predispose affected families to hereditary cancer syndromes, affording an opportunity to identify genetic lesions that also cause the more common sporadic cancers.

Prostate cancer (PRCA) is the most common cancer diagnosed (1999 estimate 179,300 cases) and the second leading cause of cancer mortality (1999 estimate 37,000 deaths) in men in the United States. Family history is the single strongest risk factor currently known for prostate cancer. This raises the possibility that heritable genetic factors may be involved in the development of this disease in a subset of men. The genetic contribution to diseases of complex origin such as cancer is often most salient in families of early onset cases. Therefore, prostate cancer inheritance following a simple Mendelian pattern, may be identified in the families of probands with early-onset cases. Common susceptibility alleles of small effect may be detectable in families with later-onset and/or less strong family history of PRCA or in case-control data.

ELIGIBILITY:
* INCLUSION CRITERIA:

Enrollment in this study includes case-control data from men with prostate cancer and matched controls who are free from the disease, plus affected and unaffected individuals from families who meet the following criteria for Hereditary Prostate Cancer:

1. A cluster of 3 or more first degree relatives, such as a father and 2 sons or 3 brothers
2. The occurrence of prostate cancer in each of 3 generations in either the proband's paternal or maternal lineages
3. Two first or second-degree relatives affected at an early age (age 55 years or younger).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing specimens
Sampling Method: Non-Probability Sample
Enrollment: 7776 (Actual)
Dates: Start 1995-01-01 (Actual); Primary Completion 2009-07-17 (Actual); Study Completion 2009-07-17 (Actual)

PRIMARY OUTCOMES:
A | Ongoing
  To identify by genetic mapping the existence of loci responsible for hereditary prostate cancer.
B | Ongoing
  To identify and characterize the gene(s) within the identified regions above, which are involved in the etiology of hereditary prostatecancer.
C | Ongoing
  To study the role of the above gene(s) in the initiation or progression of prostatic neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bailey-Wilson, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (8):
- United States (7):
  - Translational Genomics Research Institute, Phoenix, Arizona
  - Howard University Hospital, Washington D.C., District of Columbia
  - Louisiana State University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest University, Winston-Salem, North Carolina
- Tampere University, Tampere, Finland

REFERENCES:
- [Background] Ichikawa T, Ichikawa Y, Dong J, Hawkins AL, Griffin CA, Isaacs WB, Oshimura M, Barrett JC, Isaacs JT. Localization of metastasis suppressor gene(s) for prostatic cancer to the short arm of human chromosome 11. Cancer Res. 1992 Jun 15;52(12):3486-90. PMID 1596907
- [Background] Bishop JM. The molecular genetics of cancer. Science. 1987 Jan 16;235(4786):305-11. doi: 10.1126/science.3541204.
- [Background] Knudson AG Jr. Hereditary cancer, oncogenes, and antioncogenes. Cancer Res. 1985 Apr;45(4):1437-43. No abstract available. PMID 2983882
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1995-HG-0158.html